CLINICAL TRIAL: NCT03117751
Title: Total Therapy XVII for Newly Diagnosed Patients With Acute Lymphoblastic Leukemia and Lymphoma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Incyte Corporation (Industry); Amgen (Industry); Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOT17; NCI-2017-00582 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2017-03-27; First posted 2017-04-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Lymphoblastic Lymphoma
Keywords: Leukemia; Lymphoma; Pediatric; B-Cell; T-Cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphoma | interventions — Prednisone; Prednisolone; prednisolone phosphate; Vincristine; Daunorubicin; pegaspargase; Asparaginase; asparaginase erwinia chrysanthemi recombinant; Cyclophosphamide; Cytarabine; Mercaptopurine; Dasatinib; Methotrexate; blinatumomab; ruxolitinib; Bortezomib; Dexamethasone; Calcium Dobesilate; Doxorubicin; Etoposide; etoposide phosphate; Clofarabine; Vorinostat; Idarubicin; nelarabine; Thioguanine; calaspargase pegol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only certain outcome measures as indicated will be blinded to the outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- B-ALL and B-LLy, Low-risk (Experimental): Patients with low-risk B ALL and LLy will have Induction (6 weeks), Consolidation (8 weeks), and Continuation (120 weeks). During Remission Induction therapy, prednisone dose is 40mg/m^2 and 1-2 doses of daunorubicin (based on day 8 peripheral blood MRD in patients with ETV6-RUNX1 or hyperdiploid) are given. Dasatinib is given for patients with ABL-class fusion. Blinatumomab will be given to patients with certain genetic subtypes and those with Down syndrome.
  Interventions: Prednisone, vincristine, daunorubicin, pegaspargase (or Erwinase®, Rylaze™ or Calaspargase pegol), cyclophosphamide, cytarabine, mercaptopurine, dasatinib, thioguanine, methotrexate, dexamethasone, blinatumomab.
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Daunorubicin; Drug: Pegaspargase; Drug: Erwinase®; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Dasatinib; Drug: Methotrexate; Drug: Blinatumomab; Drug: Dexamethasone; Drug: Thioguanine; Drug: Asparaginase Erwinia chrysanthemi (recombinant)-rywn; Drug: Calaspargase Pegol
- B-ALL and B-LLy, Standard-risk (Experimental): Induction (6wks), Early Intensification (4wks), Consolidation (8wks) and Continuation (120 wks). Remission Induction: Prednisone dose is 40mg/m^2 and 2 doses daunorubicin are given. Dasatinib: given for patients with Ph+ and those with ABL-class fusion. Ruxolitinib: given for patients with activation of JAK-STAT signaling; ALL patients with Day 15 or Day 22 MRD ≥5%, LLy patients who don't qualify for complete response at end of Remission Induction and all patients with ETP and T/M MPAL. Bortezomib is given to patients without targetable lesions and Day 15 or Day 22 MRD >5%. Blinatumomab will be given to patients with residual disease at the end of induction (≥0.01% and <1%), certain genetic subtypes and Down syndrome.
  Interventions: prednisone, vincristine, daunorubicin, pegaspargase (or Erwinase®, Rylaze™ or Calaspargase pegol), cyclophosphamide, cytarabine, mercaptopurine, dasatinib, bortezomib, ruxolitinib, blinatumomab, thioguanine, methotrexate, dexamethasone, doxorubicin
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Daunorubicin; Drug: Pegaspargase; Drug: Erwinase®; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Dasatinib; Drug: Methotrexate; Drug: Blinatumomab; Drug: Ruxolitinib; Drug: Bortezomib; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Thioguanine; Drug: Asparaginase Erwinia chrysanthemi (recombinant)-rywn; Drug: Calaspargase Pegol
- B-ALL and B-LLy, High-risk (Experimental): Induction (6 weeks), Early Intensification (4 weeks), Consolidation (8 weeks), and Immunotherapy (chimeric antigen receptor [CAR] T cells). Patients who do not respond to Immunotherapy will receive Reintensification therapy. During Remission Induction therapy, prednisone dose is 40mg/m^2 and 2 doses of daunorubicin are given. Dasatinib, ruxolitinib, and bortezomib are given as done for patients with standard-risk B-ALL but are discontinued in Immunotherapy and Reintensification therapy. Blinatumomab will be given to patients who are not able to receive CAR T cell therapy and patients with certain genetic subtypes and those with Down syndrome.
  Interventions: prednisone, vincristine, daunorubicin, pegaspargase (or Erwinase®, Rylaze™ or Calaspargase pegol), cyclophosphamide, cytarabine, mercaptopurine, dasatinib, bortezomib, ruxolitinib, blinatumomab, etoposide, dexamethasone, clofarabine, thioguanine, methotrexate.
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Daunorubicin; Drug: Pegaspargase; Drug: Erwinase®; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Dasatinib; Drug: Methotrexate; Drug: Blinatumomab; Drug: Ruxolitinib; Drug: Bortezomib; Drug: Dexamethasone; Drug: Etoposide; Drug: Clofarabine; Drug: Thioguanine; Drug: Asparaginase Erwinia chrysanthemi (recombinant)-rywn; Drug: Calaspargase Pegol
- T-ALL and T-LLy, Standard-risk (Experimental): Induction (6 wks), Early Intensification (4 wks), Consolidation (8 wks), and Continuation (120 wks). During Remission Induction therapy, prednisone dose is 60mg/m^2 and 3 doses daunorubicin are given. Dasatinib is given for patients with Ph+ and those with ABL-class fusion. Ruxolitinib is given for patients with activation of JAK-STAT signaling; ALL patients with Day 15 or Day 22 MRD ≥5% and all patients with ETP and T/M MPAL and LLy patients who don't qualify for complete response at end of Remission Induction. Bortezomib is given to patients without targetable lesions and Day 15 or Day 22 MRD ≥ 5%.
  Interventions: prednisone, vincristine, daunorubicin, pegaspargase (or Erwinase®, Rylaze™ or Calaspargase pegol), cyclophosphamide, cytarabine, mercaptopurine, dasatinib, bortezomib, ruxolitinib, methotrexate, dexamethasone, doxorubicin, nelarabine, thioguanine.
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Daunorubicin; Drug: Pegaspargase; Drug: Erwinase®; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Dasatinib; Drug: Methotrexate; Drug: Ruxolitinib; Drug: Bortezomib; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Nelarabine; Drug: Thioguanine; Drug: Asparaginase Erwinia chrysanthemi (recombinant)-rywn; Drug: Calaspargase Pegol
- T-ALL and T-LLy, High-risk (Experimental): Induction (6 wks), Early Intensification (4 wks), Consolidation (8 wks), and Reintensification. During Remission Induction therapy, prednisone dose is 60mg/m^2 and 3 doses daunorubicin are given. Dasatinib, ruxolitinib, and bortezomib given as done for patients with standard-risk T-ALL but are discontinued in Reintensification therapy.
  Interventions: prednisone, vincristine, daunorubicin, pegaspargase (or Erwinase®, Rylaze™ or Calaspargase pegol), cyclophosphamide, cytarabine, mercaptopurine, dasatinib, bortezomib, ruxolitinib, methotrexate, etoposide, dexamethasone, clofarabine, vorinostat, idarubicin, nelarabine, thioguanine..
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Daunorubicin; Drug: Pegaspargase; Drug: Erwinase®; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Dasatinib; Drug: Methotrexate; Drug: Ruxolitinib; Drug: Bortezomib; Drug: Dexamethasone; Drug: Etoposide; Drug: Clofarabine; Drug: Vorinostat; Drug: Idarubicin; Drug: Nelarabine; Drug: Thioguanine; Drug: Asparaginase Erwinia chrysanthemi (recombinant)-rywn; Drug: Calaspargase Pegol
- ALL, CEP72 T/T, Vincristine (Experimental): Patients with the CEP72 rs904627T/T genotype (~16% of patients) will be randomized (unblinded design, only those who evaluate neuropathy are blinded) to receive either 1.5 mg/m^2 or 1 mg/m^2 of vincristine after Continuation Week 1. Patients in low- risk will complete vincristine in Week 49 and those in standard/high-risk will complete in Week 101.
  Intervention: vincristine.
  Interventions: Drug: Vincristine
- ALL, CEP72 C/T or C/C, Vincristine (Experimental): Patients with either a CEP72 rs904627 C/T or C/C genotype (~84% of patients) will be randomized (unblinded design, only those who evaluate neuropathy are blinded) to receive vincristine (2 mg/m^2 per dose except during Reinduction I and Reinduction II when 3 weekly doses of 1.5 mg/m^2 will be given) and dexamethasone pulses through Week 49 of Continuation Treatment or through Week 101 of Continuation Treatment. Patients at low-risk will complete vincristine in Week 49.
  Interventions: vincristine, dexamethasone, methotrexate, mercaptopurine.
  Interventions: Drug: Vincristine; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Dexamethasone

INTERVENTIONS:
Drug: Prednisone — Given orally (PO).
  Other Names: Prednisolone; Deltasone; Meticorten; Orasone®; Liquid Pred; Pediapred®; Sterapred®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Vincristine — Given intravenously (IV).
  Other Names: Vincristine sulfate; Oncovin®; VCR; LCR
Drug: Daunorubicin — Given IV.
  Other Names: Daunomycin; rubidomycin; Cerubidine®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Pegaspargase — Given IV or intramuscularly (IM) .
  Other Names: PEG-asparaginase; PEGLA; PEG-L-asparaginase; polyethylene glycol-L-asparaginase; Oncaspar®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Erwinase® — To be used in case of hypersensitivity or intolerance to Pegaspargase or if Pegaspargase is not available. Given IV or intramuscularly (IM).
  Other Names: Erwinia chrysanthemi; Asparaginase Erwinia chrysanthemi; Erwinaze^TM; Crisantaspase
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Cyclophosphamide — Given IV.
  Other Names: Cytoxan®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Cytarabine — Given IV or by subcutaneous injection (SQ).
  Other Names: Cytosine arabinoside; Ara-C; Cytosar®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Mercaptopurine — Given PO.
  Other Names: 6-MP; Purinethol®; Purixan^TM; 6-mercaptopurine
  Arms: ALL, CEP72 C/T or C/C, Vincristine; B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Dasatinib — Given PO.
  Other Names: Sprycel®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Methotrexate — Given IV.
  Other Names: MTX; amethopterin; Trexall®
  Arms: ALL, CEP72 C/T or C/C, Vincristine; B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Blinatumomab — Given IV.
  Other Names: Blincyto®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk
Drug: Ruxolitinib — Given PO.
  Other Names: Jakafi®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Bortezomib — Given IV or subcutaneously (SQ).
  Other Names: Velcade®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Dexamethasone — Given PO.
  Other Names: Decadron®; Hexadrol®; Dexone®; Dexameth®
  Arms: ALL, CEP72 C/T or C/C, Vincristine; B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Doxorubicin — Given IV.
  Other Names: Adriamycin®
  Arms: B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, Standard-risk
Drug: Etoposide — Given IV.
  Other Names: Etoposide Phosphate; VePesid®; Etopophos®; VP-16
  Arms: B-ALL and B-LLy, High-risk; T-ALL and T-LLy, High-risk
Drug: Clofarabine — Given IV.
  Other Names: Clolar®
  Arms: B-ALL and B-LLy, High-risk; T-ALL and T-LLy, High-risk
Drug: Vorinostat — Given PO.
  Other Names: Zolinza®; Suberoylanilide Hydroxamic Acid; SAHA
  Arms: T-ALL and T-LLy, High-risk
Drug: Idarubicin — Given IV.
  Other Names: Idarubicin HCl; 4-Demethoxydaunorubicin; 4-DMD; DMDR; Idamycin PFS®
  Arms: T-ALL and T-LLy, High-risk
Drug: Nelarabine — Given IV.
  Other Names: Arranon®; Atriance®; Compound 506U78
  Arms: T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Thioguanine — Participants with mercaptopurine-related pancreatitis. Given PO.
  Other Names: 6-thioguanine; Tioguanine; 2-amino-1,7-dihydro-6H-purine-6-thione; WR-1141; Tabloid®; Lanvis®
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Asparaginase Erwinia chrysanthemi (recombinant)-rywn — To be used in case of hypersensitivity or intolerance to Pegaspargase or if Pegaspargase is not available. Given intramuscularly (IM).
  Other Names: Rylaze™; Recombinant Erwinia
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk
Drug: Calaspargase Pegol — To be used in case of hypersensitivity or intolerance to Pegaspargase or if Pegaspargase is not available. Given IV.
  Other Names: ASPARLAS
  Arms: B-ALL and B-LLy, High-risk; B-ALL and B-LLy, Low-risk; B-ALL and B-LLy, Standard-risk; T-ALL and T-LLy, High-risk; T-ALL and T-LLy, Standard-risk

SUMMARY:
The overarching objective of this study is to use novel precision medicine strategies based on inherited and acquired leukemia-specific genomic features and targeted treatment approaches to improve the cure rate and quality of life of children with acute lymphoblastic leukemia (ALL) and acute lymphoblastic lymphoma (LLy).

Primary Therapeutic Objectives:

* To improve the event-free survival of provisional standard- or high-risk patients with genetically or immunologically targetable lesions or minimal residual disease (MRD) ≥ 5% at Day 15 or Day 22 or ≥1% at the end of Remission Induction, by the addition of molecular and immunotherapeutic approaches including tyrosine kinase inhibitors or chimeric antigen receptor (CAR) T cell / blinatumomab for refractory B-acute lymphoblastic leukemia (B-ALL) or B-lymphoblastic lymphoma (B-LLy), and the proteasome inhibitor bortezomib for those lacking targetable lesions.
* To improve overall treatment outcome of T acute lymphoblastic leukemia (T-ALL) and T-lymphoblastic lymphoma (T-LLy) by optimizing pegaspargase and cyclophosphamide treatment and by the addition of new agents in patients with targetable genomic abnormalities (e.g., activated tyrosine kinases or JAK/STAT mutations) or by the addition of bortezomib for those who have a poor early response to treatment but no targetable lesions, and by administering nelarabine to T-ALL and T-LLy patients with leukemia/lymphoma cells in cerebrospinal fluid at diagnosis or MRD ≥0.01% at the end of induction.
* To determine in a randomized study design whether the incidence and/or severity of acute vincristine-induced peripheral neuropathy can be reduced by decreasing the dosage of vincristine in patients with the high-risk CEP72 TT genotype or by shortening the duration of vincristine therapy in standard/high-risk patients with the CEP72 CC or CT genotype.

Secondary Therapeutic Objectives:

* To estimate the event-free survival and overall survival of children with ALL and to assess the non-inferiority of TOTXVII compared to the historical control given by TOTXVI.
* To estimate the event-free survival and overall survival of children with LLy when ALL diagnostic and treatment approaches are used.
* To evaluate the efficacy of blinatumomab in B-ALL patients with end of induction MRD ≥0.01% to <1% and those (regardless of MRD level or TOTXVII risk category) with the genetic subtypes of BCR-ABL1, ABL-class fusion, JAK-STAT activating mutation, hypodiploid, iAMP21, ETV6-RUNX1-like, MEF2D, TCF3-HLF, or BCL2/MYC or with Down syndrome, by comparing event-free survival to historical control from TOTXVI.
* To determine the tolerability of combination therapy with ruxolitinib and Early Intensification therapy in patients with activation of JAK-STAT signaling that can be inhibited by ruxolitinib and Day 15 or Day 22 MRD ≥5%, Day 42 MRD ≥1%, or LLy patients without complete response at the End of Induction and all patients with early T cell precursor leukemia.

Biological Objectives:

* To use data from clinical genomic sequencing of diagnosis, germline/remission and MRD samples to guide therapy, including incorporation of targeted agents and institution of genetic counseling and cancer surveillance.
* To evaluate and implement deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) sequencing-based methods to monitor levels of MRD in bone marrow, blood, and cerebrospinal fluid.
* To assess clonal diversity and evolution of pre-leukemic and leukemic populations using DNA variant detection and single-cell genomic analyses in a non-clinical, research setting.
* To identify germline or somatic genomic variants associated with drug resistance of ALL cells to conventional and newer targeted anti-leukemic agents in a non-clinical, research setting.
* To compare drug sensitivity of ALL cells from diagnosis to relapse in vitro and in vivo and determine if acquired resistance to specific agents is related to specific somatic genome variants that are not detected or found in only a minor clone at initial diagnosis.

Supportive Care Objectives

* To conduct serial neurocognitive monitoring of patients to investigate the neurocognitive trajectory, mechanisms, and risk factors.
* To evaluate the impact of low-magnitude high frequency mechanical stimulation on bone mineral density and markers of bone turnover.

There are several Exploratory Objectives.

DETAILED DESCRIPTION:
Participants will be classified into one of three categories (low-, standard-, or high-risk) based on the presenting age, leukocyte count/lymphoma staging, presence or absence of CNS-3 status or testicular disease, immunophenotype, molecular genetics, DNA index, and early response to therapy.

Treatment will consist of three main phases: Remission Induction, Consolidation, and Continuation. Early Intensification therapy will be given prior to Consolidation to patients with provisional standard-risk or high-risk ALL/LLy or any provisional low-risk patients with Day 15 MRD ≥1% as well as provisional low-risk LLy patients who do not obtain complete response at the end of Induction. Patients with mixed phenotype acute leukemia (MPAL) are treated by using the same treatment stratification used in ALL although analysis is performed separately from ALL or LLy cohorts.

Brief outline of treatment plan:

Patients will be assigned to treatment based on risk group: Low-Risk, Standard-Risk and High-Risk and cell type (T or B cell).

Remission Induction initially consists of prednisone (28 days), vincristine (4 weekly doses), daunorubicin (1 to 3 weekly doses), and pegaspargase 1 dose for all patients and 2 doses for those with Day 15 MRD 1% or higher. The second part (given over 2 weeks and overlapping with the last week of the first part of induction) consists of cyclophosphamide, cytarabine, and mercaptopurine combinations. Dasatinib will be added for patients with Ph+ and Ph-like ABL-class fusions and bortezomib will be given to patients with no targetable lesions and Day 15 or Day 22 minimal residual disease (MRD) ≥ 5% on Days 29 and 32.

Early Intensification will be given prior to Consolidation to patients with provisional standard-risk or high-risk ALL/LLy or any provisional low-risk patients with Day 15 MRD ≥1% as well as provisional low-risk LLy patients who do not obtain complete response at the end of Induction. For patients with Ph-like ALL that is targetable with JAK inhibitor and Day 15 or Day 22 MRD level ≥5% or end of Remission Induction ≥1% as well as all patients with early T cell precursor (ETP) ALL and T/M MPAL, ruxolitinib will be used. This includes, but is not limited to CRLF2, JAK2, and EPOR rearrangements and sequence/structural changes in JAK1/2, TYK2, IL7R, and SH2B3. Ruxolitinib will be added in LLy patients with activation of JAK-STAT signaling that can be inhibited by ruxolitinib whose responses do not qualify complete response at the end of Remission Induction. Dasatinib will continue for patients with ABL-class fusions. Bortezomib will be added for patients with no targetable lesions and Day 15 or Day 22 MRD ≥ 5% or LLy patients without complete response at the End of Induction.

Consolidation Treatment will consist of high dose methotrexate (HDMTX) (every other week for 4 doses); daily mercaptopurine and IT chemotherapy on the same dates of HDMTX. Dasatinib will continue for patients with ABL-class fusions. Ruxolitinib will continue for patients with activation of JAK-STAT signaling that can be inhibited by ruxolitinib and Day 15 or Day 22 MRD ≥5% or Day 42 MRD ≥1% (or for LLy patients who do not qualify complete response at the end of Remission Induction) and all cases with ETP ALL and T/M MPAL.

Immunotherapy: CAR T-cell therapy will be considered for High-risk B-ALL and B-LLy patients. Blinatumomab will be given to patients with Standard-risk B-ALL and B-LLy with residual disease at the end of induction and High-risk B-ALL and B-LLy patients who are not able to receive CAR T-cell therapy. Blinatumomab is also given to patients with the following genetic subtypes (BCR-ABL1, ABL-class fusion, JAK-STAT activating mutation, hypodiploid, iAMP21, ETV6-RUNX1-like, MEF2D, TCF3/HLF, or BCL2/MYC) or with Down syndrome, regardless of MRD level and/or Total 17 risk category.

Reintensification therapy will be offered to certain High-risk patients with persistent MRD after Immunotherapy (B-ALL and B-LLy) or Early Intensification (T-ALL and T-LLy), or those who cannot receive Immunotherapy.

Continuation Treatment will consist of 120 weeks of risk-directed therapy. Dasatinib will continue in patients with ABL-class fusion. Ruxolitinib will continue in patients with activation of JAK-STAT signaling that can be inhibited by ruxolitinib and Day 15 or Day 22 MRD ≥5% or Day 42 MRD ≥1% (or for LLy patients who do not qualify complete response at the end of Remission Induction) and all cases with ETP ALL. T-ALL and T-LLy patients with leukemia/lymphoma cells in cerebrospinal fluid at diagnosis or MRD ≥0.01% at the end of Induction will receive nelarabine. ALL/LLy Patients with the CEP72 rs904627T/T genotype (16% of patients) will be randomized (unblinded design except those who evaluate neuropathies) to receive either 1.5 mg/m2 or 1 mg/m2 of vincristine after Continuation Week 1. Patients in low- risk will complete vincristine in Week 49 and those in standard/high-risk will complete in Week 101. Standard/high-risk patients with either a CEP72 rs904627 C/T or C/C genotype (84% of patients) will be randomized to receive vincristine and dexamethasone pulses through Week 49 of Continuation Treatment or through Week 101 of Continuation Treatment. Low-risk patients will complete vincristine in Week 49.

Intrathecal therapy is given throughout the treatment. The number of intrathecal therapy is based on the risk factors of central nervous system relapse.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B- or T-ALL or LLy by immunophenotyping:
* LLy participants must have < 25% tumor cells in bone marrow and peripheral blood by morphology and flow cytometry. If any of these show ≥25% blasts, patient will be considered to have leukemia. Patients with MPAL are eligible.
* Age 1-18 years (inclusive).
* No prior therapy, or limited prior therapy, including systemic glucocorticoids for one week or less, one dose of vincristine, emergency radiation therapy (e.g., to the mediastinum, head and neck, orbit, etc.) and one dose of intrathecal chemotherapy.
* Written, informed consent and assent following Institutional Review Board (IRB), National Cancer Institute (NCI), Food and Drug Administration (FDA), and Office of Human Research Protections (OHRP) Guidelines.

Exclusion Criteria:

* Participants who are pregnant or lactating. Males or females of reproductive potential must agree to use effective contraception for the duration of study participation.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 790 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival of ALL patients (EFS) | At 3.5 years after enrollment of the last participant
  5-year EFS: Kaplan-Meier estimates of EFS curve of ALL patients will be computed and compared historically with those of the St. Jude Children's Research Hospital's (SJCRH) TOTXVI study (NCT00549848). All eligible patients entered on the current TOT17 study will be included in these comparisons. Comparisons by log-rank tests will be made both un-stratified and stratified by risk groups.
Proportion of patients with CEP72TT genotype who develop two or more episodes of Grade 2 or higher neuropathy during Continuation | At 6 months after the last randomized patient completes Continuation Treatment (Week 120).
  This will be a single-blind, stratified block randomized experiment. Although the investigators who evaluate neuropathy and neuropathic pain and the patients are blinded for treatment assignment, treating clinicians and pharmacy staff are not. Patients will be randomized at a 1:1 ratio into two treatment groups: 1.5 mg/m^2 vs. 1 mg/m^2 vincristine (VCR) dose. Randomization will be stratified by two factors known to significantly affect neuropathy during the Continuation phase, namely, Grade 2 or higher neuropathy prior to Continuation (none, 1 episode, 2 or more episodes) and race (black, others). The proportion of patients who develop two or more episodes of Grade 2 or higher neuropathy during Continuation Treatment will be compared between the two VCR dose groups, using a Z-test for two sample proportions.
Cumulative incidence of Grade 2 or higher neuropathy in patients with CEP72 CC or CT genotype | After the last randomized patient is followed for 1 year after Week 101 of Continuation therapy
  This will be a single blind stratified block randomized experiment. The investigators who evaluate neuropathy and neuropathic pain and the patients are blinded for treatment assignment. Treating clinicians and pharmacy staff will not be blinded. Standard/high-risk patients will be randomized at a 1:1 ratio into two treatment groups at Week 49 of Continuation therapy: to vincristine + dexamethasone (VCR+DEX) pulses or to 6-mercaptopurine + methotrexate (6MP+MTX). The primary analysis will compare the cumulative incidence of the first episode of Grade 2 or higher neuropathy or neuropathic pain (the end point) by stratified Gray's test. Adverse events other than the endpoint rendering a patient drop out after Continuation Week 49 are regarded as competing events.

SECONDARY OUTCOMES:
5-year overall survival (OS) of ALL patients compared to historical controls | 3.5 years after enrollment of the last patient
  Kaplan-Meier estimates of OS curve of ALL patients will be computed and compared historically with those of the St. Jude Children's Research Hospital's (SJCRH) TOTXVI study (NCT00549848). All eligible patients entered on the current TOT17 study will be included in these comparisons. Comparisons by log-rank tests will be made both un-stratified and stratified by risk groups.
EFS of LLy patients | 3.5 years after enrollment of the last patient
  5-year EFS: Kaplan-Meier estimates of EFS curve in patients with LLy will be computed.
5-year OS of LLy patients | 3.5 years after enrollment of the last patient
  Kaplan-Meier estimates of OS curve in patients with LLy will be computed.
The efficacy of blinatumomab in B-ALL patients | 3.5 years after enrollment of the last patient
  Comparison with historical control by log-rank tests will be performed.
Comparison of MRD measurements between flow cytometry and sequencing | From Day 8 through Day 42 after remission induction (At 6 months after enrollment of the 40^t^h evaluable patient)
  For this comparison, 40 patients will be accrued for Day 8, Day 15 and Day 42 MRD, and primarily assess the correlation and concordance between the two methods at these time points if sufficient cells are available, and secondarily analyze for Day 22 and MRD levels obtained after remission induction.
Log hazard ratio of the association of low level of MRD and treatment outcome | 3.5 years after enrollment of the last patient
  The investigators will analyze the association of next-generation sequencing-determined MRD level (as a continuous variable) with the risk of relapses in bone marrow and possibly other sites (bone marrow or combined relapses). Fine-Gray regression model will be applied to estimate the hazard ratio of relapse as a function of the increase in MRD level.
Comparison of bone marrow and peripheral blood MRD | From Day 15 through Day 42 of remission induction and end of therapy (At 6 months after enrollment of the last evaluable patient)
  Parametric (linear) or non-parametric (if necessary) regression models will be fitted to analyze the relationship between the MRD levels in peripheral blood by sequencing methods and MRD levels in bone marrow (by sequencing or flow cytometry). The peripheral blood MRD level corresponding to 0.01% in bone marrow is then obtained by solving the (regression) equation for the peripheral blood MRD level.
Isolated CNS relapse in CNS1b patients | 3.5 years after enrollment of the last patient
  Traditional CNS2 patients with negative TdT and negative next-generation sequencing results will receive CNS1 therapy on TOT17. Risk of isolated CNS relapse in this subset of patients will be compared to that in the CNS2 patients treated on TOTXV and TOTXVI, using stratified (by protocol) Gray's test.
Level of clonal diversity and rise of leukemic clones during treatment | From Day 1 through week 120 of continuation (at 6 months after the last enrolled patient completes Week 120)
  In this study the investigators will use single-cell, cell-free, and bulk population sequencing to monitor somatic mutations in peripheral blood as patients undergo treatment, which will be correlated with clonal diversity at diagnosis, in vitro chemotherapy resistance, MRD, and patient outcome.
Number and type of germline or somatic genomic variants associated with drug resistance | 3.5 years after enrollment of the last participant
  The number and type of germline or somatic genomic variants associated with drug resistance of ALL cells to conventional and newer targeted anti-leukemic agents in a non-clinical, research setting will be given.
Comparison of drug sensitivity of ALL cells between diagnosis and relapse in vitro and in vivo | 5 years after enrollment of the last participant
  To compare drug sensitivity of ALL cells from diagnosis to relapse in vitro and in vivo and determine if acquired resistance to specific agents is related to specific somatic genome variants that are not detected or found in only a minor clone at initial diagnosis
Change in bone mineral density (BMD) in the tibia | From baseline to week 49 Continuation treatment (up to 6 months after last patient completes week 49 Continuation)
  The primary outcome is BMD in the tibia, measured at baseline and the end of intervention. The changes from baseline to the end of the intervention between the treatment and control groups will be compared.
Change in markers of bone turnover | From baseline to week 49 Continuation treatment (up to 6 months after last patient completes week 49 Continuation)
  Linear mixed models or other methods will be used to evaluate this outcome.

OTHER OUTCOMES:
Log odds ratio of pharmacogenetic predictors of treatment outcome (host toxicity or in vivo efficacy) | 5 years after enrollment of the last participant
  The log odds ratio of pharmacogenetics predictors of treatment outcome will be given.
Log odds ratio of pharmacokinetic predictors of treatment outcome (host toxicity or in vivo efficacy) | 5 years after enrollment of the last participant
  The log odds ratio of pharmacokinetic predictors of treatment outcome will be given.
Log odds ratio of pharmacodynamic predictors of treatment outcome (host toxicity or in vivo efficacy) | 5 years after enrollment of the last participant
  The log odds ratio of pharmacodynamic predictors of treatment outcome will be given.
Thiopurine metabolism | 3.5 years after enrollment of the last participant
  A detailed assessment of thiopurine metabolism will be done and correlated with 6-mercaptopurine (6MP) tolerance, toxicity, and treatment outcome.
Number of participants experiencing specific therapy-related infection events | 1 year after completion of therapy for last enrolled patient (up to 3.5 years after enrollment)
  All enrolled participants will be eligible for this component. Descriptive statistics, such as frequency and proportion, will be summarized for breakthrough infections, antibiotic-resistant infections, febrile neutropenia episodes and adverse events. Cumulative incidence of breakthrough infection, febrile neutropenia and adverse events will also be explored, with competing risks and/or recurrent event appropriately adjusted.
5-year EFS of MPAL patients | 3.5 years after enrollment of the last patient
  Kaplan-Meier estimates of EFS curve in patients with MPAL will be computed.
5-year OS of MPAL patients | 3.5 years after enrollment of the last patient
  Kaplan-Meier estimates of OS curve in patients with MPAL will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroto Inaba, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (8):
- United States (7):
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital of Illinois at OSF-Saint Francis Medical Center (St. Jude Midwest Affiliate - Peoria), Peoria, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. Jude Affiliate Clinic - Novant Health Hemby Children's Hospital, Charlotte, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
- The Royal Children's Hospital Melbourne, Parkville, Victoria, Australia

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT03117751/ICF_000.pdf